CLINICAL TRIAL: NCT05238675
Title: A Randomised, Double-blind, Placebo-controlled, Parallel Group, Dose-finding Study Evaluating Efficacy, Safety and Tolerability of BI 1291583 qd Over at Least 24 Weeks in Patients With Bronchiectasis (AirleafTM)
Brief Title: A Study to Test Whether Different Doses of BI 1291583 Help People With Bronchiectasis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1397-0012; 2021-003304-41 (EudraCT Number)
Record Dates: First submitted 2022-02-03; First posted 2022-02-14 (Actual); Last update posted 2025-08-14 (Actual); Status verified 2025-08

CONDITIONS: Bronchiectasis
MeSH Terms: conditions — Bronchiectasis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- BI 1291583: Low dose group (Experimental)
  Interventions: Drug: BI 1291583
- BI 1291583: Medium dose group (Experimental)
  Interventions: Drug: BI 1291583
- BI 1291583: High dose group (Experimental)
  Interventions: Drug: BI 1291583
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: BI 1291583 — BI 1291583
  Other Names: Verducatib
  Arms: BI 1291583: High dose group; BI 1291583: Low dose group; BI 1291583: Medium dose group
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
This study is open to adults with bronchiectasis. People can join the study if they produce sputum and have a history of flare-ups (also called exacerbations).

The purpose of this study is to find out whether a medicine called BI 1291583 helps people with bronchiectasis.

Participants are put into 4 groups randomly, which means by chance. Participants in groups 1, 2, and 3 get different doses of BI 1291583. Participants in group 4 get placebo. Placebo tablets look like BI 1291583 tablets, but do not contain any medicine. Participants take the tablets once a day.

Participants are in the study for between 6 months and 1 year. During this time, they visit the study site about 10 times and get about 5 phone calls from the site staff.

The doctors document when participants experience flare-ups during the study. The time to the first flare-ups is compared between the treatment groups. Doctors also regularly check participants' health and take note of any unwanted effects.

ELIGIBILITY:
Inclusion Criteria:

- Male or female patients: Women of childbearing potential (WOCBP) must be ready and able to use highly effective methods of birth control per ICH M3 (R2) that result in a low failure rate of less than 1% per year when used consistently and correctly, as well as one barrier method. A list of contraception methods meeting these criteria is provided in the patient information.

Men participating in this clinical trial must use male contraception (condom or sexual abstinence) if their sexual partner is a WOCBP.

* Signed and dated written informed consent prior to admission to the study, in accordance with Good Clinical Practice (GCP) and local legislation.
* Age of patients when signing the informed consent ≥18 (for Korea: ≥19) and ≤85 years.
* Clinical history consistent with bronchiectasis (e.g., cough, chronic sputum production and/or recurrent respiratory infections) and investigator confirmed diagnosis of bronchiectasis by computed tomography (CT) scan. Subjects whose past chest radiographic image records are not available will undergo a chest CT scan during Screening. Historical scans must not be older than 5 years.
* History of pulmonary exacerbations requiring antibiotic treatment. In the 12 months before Visit 1, patients must have had either:

  * at least 2 exacerbations, or
  * at least 1 exacerbation and a St. George´s Respiratory Questionnaire (SGRQ) Symptoms score of >40 at screening visit 1.

For patients on stable oral or inhaled antibiotics as chronic treatment for bronchiectasis, at least one exacerbation must have occurred since initiation of stable antibiotics.

- Current sputum producers with a history of chronic expectoration who are able to provide a spontaneous (not induced) sputum sample at Screening Visit 1.

Exclusion Criteria:

Laboratory and medical examination

* Aspartate Aminotransferase (AST) and / or Alanine Aminotransferase (ALT) >3.0 x upper limit of normal (ULN) at Visit 1, or moderate or severe liver disease (defined by Child-Pugh score B or C hepatic impairment).
* Estimated glomerular filtration rate (eGFR) according to Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) formula < 30 mL/min at Visit 1.
* An absolute blood neutrophil count <1,000/mm^3 at Visit 1 (equivalent to <1,000 cells/µL or <109 cells/L).
* Any findings in the medical examination and/or laboratory value assessed at Screening Visit 1 or during screening period, that in the opinion of the investigator may put the patient at risk by participating in the trial.
* Positive serological tests for hepatitis B, hepatitis C, or human immunodeficiency virus (HIV) infection, or known infection status.

Concomitant diagnosis and therapy

* A current diagnosis of:

  * Cystic Fibrosis
  * Hypogammaglobulinemia
  * Common variable immunodeficiency
  * α1-antitrypsin deficiency being treated with augmentation therapy
  * Allergic bronchopulmonary aspergillosis being treated or requiring treatment
  * Tuberculosis or non-tuberculous mycobacterial infection being treated or requiring treatment according to local guidelines
  * Palmoplantar keratosis; or keratoderma climactericum
  * Hypothyroidism, myxedema, chronic lymphedema with associated hyperkeratosis of the skin, acrocyanosis. If a subject has hypothyroidism but is treated and compensated, the subject is allowed into the trial
  * Psoriasis affecting palms and soles; or body surface area for psoriasis ≥ 10%
  * Reactive arthritis (Reiter's syndrome); keratoderma blennorrhagicum
  * Pityriasis rubra pilaris
  * Atopic dermatitis affecting palms and soles; or body surface area for atopic dermatitis ≥ 10%
  * Active extensive verruca vulgaris, as per investigator's discretion
  * Active fungal infection of hand and/or feet not adequately treated, or not responsive to antifungal therapy, as per investigator's discretion.
* Any clinically relevant (at the discretion of the investigator) acute respiratory infection within 4 weeks prior Visit 2, or any other acute infection requiring systemic or inhaled anti-infective therapy within 4 weeks prior Visit 2.
* Any evidence of a concomitant disease, such as Papillon-Lefevre Syndrome, relevant pulmonary, gastrointestinal, hepatic, renal, cardiovascular, metabolic, immunological, hormonal disorders, or patients who are immunocompromised with a higher risk of invasive pneumococcal disease or other invasive opportunistic infections (such as histoplasmosis, listeriosis, coccidioidomycosis, pneumocystosis), that in the opinion of the investigator, may put the patient at risk by participating in the study.
* Received any live attenuated vaccine within 4 weeks prior to Visit 2.
* Medical conditions associated with periodontal disease (to be evaluated by a periodontist or dentist):

  * Any tooth that can potentially cause pain or infection as noted in the oral exam unless they are corrected before the study (e.g. pulp necrosis).
  * Severe periodontal disease defined as with pocket depth measurements ≥ 6 mm on 2 or more teeth.
  * Class-3 mobility or Class-3 furcation involvement.
  * Scheduled tooth extraction during the study period.
* Patients who must or wish to continue the intake of restricted medications or any drug considered likely to interfere with the safe conduct of the trial.

Further exclusion criteria apply

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 322 (Actual)
Dates: Start 2022-04-28 (Actual); Primary Completion 2024-05-01 (Actual); Study Completion 2024-05-30 (Actual)

PRIMARY OUTCOMES:
Time to first pulmonary exacerbation up to 48 weeks after first drug administration | Up to week 48

SECONDARY OUTCOMES:
Key secondary: Rate of pulmonary exacerbations (number of events per person-time) up to week 48 after first drug administration | Up to week 48
Absolute change from baseline in Quality of Life Questionnaire - Bronchiectasis (QOLB) respiratory symptoms domain score at week 24 after first drug administration | At baseline and at week 24
Relative change from baseline in neutrophil elastase (NE) activity in sputum at week 12 after first drug administration | At baseline and at week 12
Absolute change from baseline in St. George's Respiratory Questionnaire (SGRQ) Symptoms score at week 24 after first drug administration | At baseline and at week 24
Absolute change from baseline in percent predicted post-bronchodilator forced expiratory volume in one second (FEV1%pred) at week 24 after first drug administration | At baseline and at week 24
Occurrence of an exacerbation by week 24 after first drug administration | Up to week 24

CONTACTS AND LOCATIONS:
Locations (112):
- United States (16):
  - Phoenix Medical Group, Peoria, Arizona
  - Newport Native MD, Inc, Newport Beach, California
  - University of California Davis, Sacramento, California
  - Central Florida Pulmonary Group, Altamonte Springs, Florida
  - Malcom Randall VA Medical Center, Gainesville, Florida
  - University of Florida College of Medicine, Jacksonville, Florida
  - University of Kansas Medical Center, Kansas City, Kansas
  - New York University Langone Medical Center, New York, New York
  - NewYork-Presbyterian/Weill Cornell Medical Center, New York, New York
  - Southeastern Research Center, Winston-Salem, North Carolina
  - University of Cincinnati, Cincinnati, Ohio
  - Medical University of South Carolina, Charleston, South Carolina
  - Institute for Translational Oncology Research, Greenville, South Carolina
  - Metroplex Pulmonary & Sleep Center, McKinney, Texas
  - Diagnostics Research Group, San Antonio, Texas
  - University of Texas Health Science Center at Tyler, Tyler, Texas
- Australia (6):
  - Macquarie University, North Ryde, New South Wales
  - Westmead Hospital, Westmead, New South Wales
  - Lung Research Queensland, Chermside, Queensland
  - Mater Research Institute, South Brisbane, Queensland
  - Institute for Respiratory Health, Nedlands, Western Australia
  - Trialswest, Spearwood, Western Australia
- Belgium (2):
  - UNIV UZ Gent, Ghent
  - UZ Leuven, Leuven
- Bulgaria (5):
  - Medical Center "Zdrave-1", Kozloduy
  - Medica Center Hera - Montana Branch, Montana
  - Medical Center ReSpiro Ltd, Razgrad
  - SHATPFD "Dr. Dimitar Gramatikov", Rousse
  - Medical Center Hera EOOD, Sofia
- Canada (3):
  - Jewish General Hospital, Montreal, Migration Data
  - Centre Hospitalier de l'Universite de Montreal (CHUM), Montreal, Quebec
  - IUCPQ (Laval University), Québec
- Czechia (2):
  - Pulmonary Private Practice Kralupy, Kralupy nad Vltavou
  - The First Pulmonary Private Practice, Prague
- Denmark (6):
  - Aalborg Sygehus Syd, Aalborg
  - Hvidovre Hospital, Hvidovre
  - Copenhagen University Hospital, Rigshospitalet, København Ø
  - Odense University Hospital, Odense
  - Sjællands Universitetshospital, Roskilde
  - Vejle University Hospital, Vejle
- France (4):
  - HOP Amiens-Picardie Sud, Amiens
  - HOP Arnaud de Villeneuve, Montpellier
  - HOP Cochin, Paris
  - HOP Pontchaillou, Rennes
- Germany (9):
  - Charité - Universitätsmedizin Berlin, Berlin
  - Ruhrlandklinik, Westdeutsches Lungenzentrum am Universitätsklinikum Essen gGmbH, Essen
  - IKF Pneumologie GmbH & Co. KG, Frankfurt
  - Velocity Clinical Research Germany GmbH, Großhansdorf
  - Lungenfachklinik Immenhausen, Immenhausen
  - Klinikum Konstanz, Konstanz
  - Velocity Clinical Research Germany GmbH, Lübeck
  - Klinikum der Universität München - Campus Innenstadt, München
  - Velocity Clinical Research Germany GmbH, Wiesbaden
- Univ. Gen. Hosp. of Ioannina, Ioannina, Greece
- Hungary (2):
  - Semmelweis University, Budapest
  - Da Vinci Private Clinic, Pécs
- Israel (4):
  - Soroka Univ. Medical Center, Beersheba
  - Lady Davis Carmel Medical Center, Haifa
  - Hadassah Medical Center, Ein-Karem, Jerusalem
  - Sourasky Medical Center, Tel Aviv
- Italy (3):
  - A.O. Univ. Policlinico "Paolo Giaccone", Palermo
  - Fondazione IRCCS Policlinico S. Matteo, Pavia
  - Istituto Clinico Humanitas, Rozzano (MI)
- Japan (13):
  - Nagoya University Hospital, Aichi, Nagoya
  - Hirosaki University Hospital, Aomori, Hirosaki
  - Kameda Clinic, Chiba, Kamogawa
  - Kyushu University Hospital, Fukuoka, Fukuoka
  - Fukuoka University Hospital, Fukuoka, Fukuoka
  - Ibarakihigashi National Hospial, Ibaraki, Naka-gun
  - Kagoshima University Hospital, Kagoshima, Kagoshima
  - Matsusaka City Hospital, Mie, Matsusaka
  - Niigata University Medical and Dental Hospital, Niigata, Niigata
  - Osaka Toneyama Medical Center, Osaka, Toyonaka
  - Saga University Hospital, Saga, Saga
  - Fukujuji Hospital, Tokyo, Kiyose
  - Kitasato Institute Hospital, Tokyo, Minato-ku
- Latvia (6):
  - Daugavpils Regional Hospital LTD Centre Outpatient Clinic, Daugavpils
  - Med.Center OLVI Health Center Assotiation,Private Practice, Daugavpils
  - VCA Dubultu Medical center, Jūrmala
  - Riga 1st Hospital, Riga
  - Pauls Stradins Clinical University Hospital, Riga
  - LUMPII Doctors practice, Riga
- Mexico (6):
  - Mediadvance Clinical S.A.P.I de C.V., Chihuahua City
  - Accelerium S de RL de CV, Monterrey
  - Hospital Universitario Nuevo de Nuevo León - CEPREP, Monterrey, Nuevo León
  - Hospital Universitario Dr Jose Eleuterio Gonzalez, Nuevo León
  - Oaxaca Site Management Organization, S.C., Oaxaca City
  - Clinical Research Institute S.C., Tlalnepantla
- Netherlands (2):
  - Amsterdam UMC, location VUMC, Amsterdam
  - Gelre Ziekenhuis Zutphen, Zutphen
- Poland (5):
  - Respiratory Medicine Centre, private prac., Bialystok, Bialystok
  - Screenmed Sp. z o.o., Piaseczno
  - Alergopneuma Medical Center, Świdnik
  - Altamed Specjalistyczna Praktyka Lekarska Pawel Siwinski, Warsaw
  - Dr. Piotr Napora, Center of Clinical Research, Wroclaw
- ULS de Santa Maria, E.P.E, Lisbon, Portugal
- South Korea (5):
  - Chungbuk National University Hospital, Cheongju-si
  - Asan Medical Center, Seoul
  - Korea University Guro Hospital, Seoul
  - SMG-SNU Boramae Medical Center, Seoul
  - The Catholic University of Korea, Eunpyeong St. Mary's Hospital, Seoul
- Spain (5):
  - Hospital Clínic de Barcelona, Barcelona
  - Hospital de Bellvitge, L'Hospitalet de Llobregat
  - Hospital General Universitario Gregorio Marañón, Madrid
  - Hospital de Mérida, Mérida
  - Hospital Quirónsalud Madrid, Pozuelo de Alarcón
- Turkey (Türkiye) (3):
  - Uludag Universitesi Tip Fakultesi, Bursa
  - Marmara University Pendik Training and Research Hospital, Istanbul
  - Sureyyapasa Egitim ve Arastirma Hastanesi, Istanbul
- United Kingdom (3):
  - Royal Papworth Hospital, Cambridge
  - Ninewells Hospital & Medical School, Dundee, Scotland
  - Liverpool Heart & Chest Hospital, Liverpool

IPD SHARING:
Plan to Share IPD: Yes
After the study is completed and the primary manuscript is accepted for publishing, researchers can use this following link https://www.mystudywindow.com/msw/datasharing to request access to the clinical study documents regarding this study, and upon a signed "Document Sharing Agreement".
  Also, Researchers can use the following link http://trials.boehringeringelheim.com/ to find information in order to request access to the clinical study data, for this and other listed studies, after the submission of a research proposal and according to the terms outlined in the website.
  The data shared are the raw clinical study data sets.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: After all regulatory activities are completed in the US and EU for the product and indication, and after the primary manuscript has been accepted for publication.
Access Criteria: For study documents - upon signing of a 'Document Sharing Agreement'. For study data - 1. after the submission and approval of the research proposal (checks will be performed by both the independent review panel and the sponsor, including checking that the planned analysis does not compete with sponsor's publication plan); 2. and upon signing of a 'Data Sharing Agreement'.
URL: https://www.mystudywindow.com/msw/datasharing

REFERENCES:
- [Derived] Chalmers JD, Shteinberg M, Mall MA, O'Donnell AE, Watz H, Gupta A, Frahm E, Eleftheraki A, Rauch J, Chotirmall SH, Armstrong AW, Eickholz P, Hasegawa N, Sauter W, McShane PJ. Cathepsin C (dipeptidyl peptidase 1) inhibition in adults with bronchiectasis: AIRLEAF, a phase II randomised, double-blind, placebo-controlled, dose-finding study. Eur Respir J. 2025 Jan 2;65(1):2401551. doi: 10.1183/13993003.01551-2024. Print 2025 Jan. PMID 39255990
- See also: Related Info — http://www.mystudywindow.com